CLINICAL TRIAL: NCT01295268
Title: The Efficacy of Emu Oil vs. Placebo in Minimizing Vulvar Pain Levels in Women--A Randomized, Double Blinded, Placebo-Controlled Trial.
Brief Title: Study of Emu Oil vs. Placebo for Vulvar Pain in Women.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: enrollment volume due to placebo arm of trial
Sponsor: Corewell Health East (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2011-019
Record Dates: First submitted 2011-02-10; First posted 2011-02-14 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2012-05

CONDITIONS: Vulvodynia; Vestibulodynia
Keywords: Vulvar pain; Vulvodynia; Vestibulodynia; Vulvar vestibulitis
MeSH Terms: conditions — Vulvodynia; Vulvar Vestibulitis | interventions — emu Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Emu Oil (Active Comparator)
  Interventions: Other: Emu Oil
- inert oil (Placebo Comparator)
  Interventions: Other: Inert oil

INTERVENTIONS:
Other: Emu Oil — Subjects will apply a specified amount of emu oil daily to area.
  Arms: Emu Oil
Other: Inert oil — A specified amount of inert oil will be applied daily to area.
  Arms: inert oil

SUMMARY:
The goal of this study is to determine if vulvar (external female genitalia) pain is decreased with emu oil over a similar placebo oil (no active ingredient) by using measurement devices, examinations, and questionnaires. Topical emu oil has not been scientifically studied for this condition yet, but related reports show no significant side effects or potential benefits.

A total of 30 women will participate in the study at William Beaumont Hospital, Royal Oak.

DETAILED DESCRIPTION:
* Women of all ages with vulvar pain may participate in this trial.
* Women will be randomized into 2 groups--a treatment group or placebo group for the 1 month study.
* At the end of the study, those in the placebo group may choose to participate in a 1 month follow-up evaluation using emu oil.

ELIGIBILITY:
Inclusion Criteria:

* Women with vulvar pain upon q-tip exam of > 3/10 at 2 or more sites tested.
* Age 18 or older.
* Capable of giving informed consent.
* Capable and willing to follow all study procedures.

Exclusion Criteria:

* Pregnant women or those intending to become pregnant during the study period.
* Vaginitis (may be treated, then tested later).
* Vulvar disease (other than vulvodynia)-lichen planus, lichen sclerosis, neoplasia, tissue damage due to radiation.
* The subject is deemed unsuitable for enrollment by the investigators based on their history or physical examination.
* Neuropathy.
* Currently in pelvic floor physical therapy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2011-02; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
The change in the Global Response Assessment (GRA) for vulvar pain. | After 1 month of intervention
  Those "moderately" or "markedly" improved on the GRA are responders

SECONDARY OUTCOMES:
The change in vulvar pain levels | After 1 month of intervention
  Based on a pain visual analog scale (VAS) and vulvalgesiometer evaluations.

CONTACTS AND LOCATIONS:
Overall Officials: Donna J Carrico, WHNP, MS, Principal Investigator — Corewell Health East
Locations (1):
- Beaumont Women's Urology Center, Royal Oak, Michigan, United States